CLINICAL TRIAL: NCT01292096
Title: Intervening With and Improving Care for Patients at Risk for Frequent Hospital Admissions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: United Hospital Fund (Other); The New York Community Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 07-649
Record Dates: First submitted 2011-01-31; First posted 2011-02-09 (Estimated); Last update posted 2016-03-02 (Estimated); Status verified 2016-02

CONDITIONS: Hospitalization; Patient Readmission
Keywords: homelessness; substance use; frequent hospitalization; frequent users of health services; enhanced care management; coordination services p; high risk for frequent hospitalization
MeSH Terms: conditions — Substance-Related Disorders | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Provision of extra (care coordination and management) services — The pilot intervention begins at the patient's bedside in the hospital and continue after his/her discharge into the community, utilizing a flexible and intensive care management model with a multi-disciplinary team approach. Community Based Care Managers (CBCMs) overseen by a social worker, will connect patients to needed community services including housing for homeless patients, accompany patients to appointments and facilitate transportation to medical, benefits enrollment, and perform other services based in the hospital and community.

SUMMARY:
Patients with frequent hospital admissions account for a disproportionate share of visits and costs. An intervention that can bridge the gap between hospital and community based care for a population of patients with frequent hospital admissions may offer both improved care and cost savings if hospital admissions can be appropriately reduced. We are now using data from our previous research to inform the development and implementation of an intervention at Bellevue Hospital, which will bridge the gap between hospital and community based care for a population of patients with frequent hospital admissions.

We hypothesize that such an intervention can offer both improved care and cost savings if hospital admissions can be appropriately reduced.

In this protocol we outline a strategy to pilot a small-scale intervention on a small subset of patients admitted to an urban public tertiary care safety net hospital who are defined by our study criteria as at high risk for future readmission. By piloting components of the intervention, we aim to assure the intervention functions as planned, and can deliver the needed services to high risk patients in a seamless and patient-centered manner. The purpose of this "feasibility study" is to ensure that when our intervention is implemented on a larger scale, it appropriately serves enrolled patients needs, and that we are able to effectively follow patients during the intervention period.

DETAILED DESCRIPTION:
In pilot research, we found that high users at Bellevue Hospital Center had varied indications for admission to the hospital, but also shared many risk factors that have been traditionally difficult for the health care system to address, including homelessness, social isolation, substance use, depression and anxiety, and fragmented primary care. Coordination of the multiple service types required to improve care for such patients across hospitals, clinics, and community-based organizations is hindered by financial disincentives, restrictive funding streams, and poor communication among service providers Intervention model and team: The pilot intervention will begin at the patient's bedside in the hospital and continue after his/her discharge into the community, utilizing a flexible and intensive care management model with a multi-disciplinary team approach. Community Based Care Managers (CBCMs) overseen by a social worker, will connect patients to needed community services including housing for homeless patients, accompany patients to appointments and facilitate transportation to medical, benefits enrollment, and perform other services based in the hospital and community.

So that the intervention can address the multitude of complex medical and social needs of high risk patients, in addition to our community partners that address the needs of homeless patients, we will partner with additional community providers of mental health, substance use, and home medical services who will assist our intervention team staff in managing patients' care after hospital discharge. In addition, we will build upon existing specialized health and social services within Bellevue Hospital (e.g. provision of prompt outpatient clinic appointments) so that this population is better and more effectively served.

Specific Aims

1) evaluate the patient and provider experience with various potential components of a pilot intervention plan for high risk, high cost patients, (identified using a predictive case-finding algorithm) conducted in partnership with community providers of homeless, mental health, substance use, and other key services, and 2) evaluate the feasibility of several aspects of the intervention. By piloting and evaluating components of the intervention, we aim to assure the intervention functions as planned, and can deliver the needed services to high risk patients.

Outcomes:

Ability of intervention team to:

1. Function effectively (e.g. communicate and coordinate with one another and with other departments in the hospital)
2. Match patients to appropriate services
3. Obtain supportive housing for homeless patients with Common Ground partner
4. Maintain contact with patients after initial hospital discharge
5. Facilitate patient adherence to outpatient appointments
6. Link patients with no usual source of care to PMD

ELIGIBILITY:
Inclusion Criteria:

* Patients identified at the time of a current hospital admission by a predictive algorithm (algorithmic risk score of 50 or greater) as being at high risk for hospital readmission in the following 12 months
* English or Spanish speaking
* Fee-for-service Medicaid or uninsured patients
* Ages 18-64

Exclusion Criteria:

* Neither English or Spanish-speaking,
* Institutionalized when not admitted to the hospital
* Unable to communicate
* HIV positive (because HIV positive patients have resources available to them from different and unrelated funding streams, and receive primary care at an off-site location)

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2007-08; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Housing placement | 1 year
  Number of eligible chronically homeless patients placed in transitional or permanent housing

SECONDARY OUTCOMES:
Patient retention in program | 1 year
  Number of subjects lost to follow-up and who did not engage after program enrollment
Linkage to primary care provider | 1 year
  Number of patients without a primary care provider who were successfully linked to primary care (at least two visits)

CONTACTS AND LOCATIONS:
Locations (1):
- Bellevue Hospital Center Department of Emergency Medicine, A345, New York, New York, United States

REFERENCES:
- [Derived] Raven MC, Doran KM, Kostrowski S, Gillespie CC, Elbel BD. An intervention to improve care and reduce costs for high-risk patients with frequent hospital admissions: a pilot study. BMC Health Serv Res. 2011 Oct 13;11:270. doi: 10.1186/1472-6963-11-270. PMID 21995329